CLINICAL TRIAL: NCT03344614
Title: An Open Single Arm Exploratory Study of Apatinib Mesylate Tablets in Combination With Raltitrexed Treatment in Patients With Advanced Colorectal Cancer
Brief Title: A Study of Apatinib in Combination With Raltitrexed Treatment in Patients With Advanced Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Dai, Guanghai, Department Director,M.D., Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AHEAD-311
Record Dates: First submitted 2017-10-31; First posted 2017-11-17 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-10

CONDITIONS: Colorectal Cancer
Keywords: third-line treatment; apatinib; raltitrexed
MeSH Terms: conditions — Colorectal Neoplasms | interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- raltitrexed combined with apatinib (Experimental): therapeutic regimen : raltitrexed, 3 mg/㎡, ivgtt, d1, apatinib 500 mg, QD po, d1-21, Every 3 weeks for 1 cycles.
  Interventions: Drug: raltitrexed combined with apatinib

INTERVENTIONS:
Drug: raltitrexed combined with apatinib — raltitrexed, 3 mg/㎡, ivgtt, d1, apatinib 500 mg, QD po, d1-21, Every 3 weeks for 1 cycles

SUMMARY:
30 patients with advanced colorectal cancer will be enrolled to observe the efficacy and safety of raltitrexed combined with apatinib as a third-line treatment.

DETAILED DESCRIPTION:
In this study, we plan to enroll 30 patients with advanced colorectal cancer after failure of second-line standard chemotherapy. The therapeutic regimen is raltitrexed, 3 mg/㎡, ivgtt, d1, apatinib 500 mg, qd,po, d1-21, Every 3 weeks for 1 cycles, the primary end point was PFS, the secondary end point was OS, DCR, ORR etc. Aim to observe the efficacy and safety of raltitrexed combined with apatinib as a third-line treatment of in patients with advanced colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* 1.Male or female, ≥ 18 of age;
* 2.Histological confirmed advanced colorectal adenocarcinoma，and at least one measurable lesion;
* 3.Have failed for ≥ 2 lines of standard chemotherapy(included Fluorouracil, irinotecan and oxaliplatin);
* 4.ECOG performance status 0-2;
* 5.Life expectancy of more than 3 months;
* 6.The main organs function is well, and randomized within 14 days before the relevant inspection indicators to meet the following requirements:

  1. blood routine test Hgb ﹥90g/L, ANC﹥1.5×109/L, Platelets ﹥ 100×109/L,
  2. biochemical tests Serum Total bilirubin ≤ 1.5 X UNL(upper normal limit), ALT or AST ≤ 2 xUNL, and ﹤ 5 x UNL（Hematogenous metastases）, Creatinine clearance rate≥ 60 ml/min(Cockcroft-Gault formula),
  3. Doppler echocardiography assessment：LVEF ≥ 50%;
* 7.No serious heart, lung, liver, kidney dysfunction; no jaundice and gastrointestinal obstruction; no acute infection;
* 8.Signed informed consent;
* 9.Good compliance, and family members agree to receive survival follow-up.

Exclusion Criteria:

* 1.Factors that could have an effect on oral medication (such as inability to swallow, chronic diarrhea and intestinal obstruction);

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-01-01 (Estimated); Study Completion 2019-07-01 (Estimated)

PRIMARY OUTCOMES:
PFS | 6 months
  Progression-free survival progression-free survival

SECONDARY OUTCOMES:
OS | 12 months
  overall survival
ORR | 12 months
  Objective Response Rate
DCR | 12 months
  Disease Control Rate

CONTACTS AND LOCATIONS:
Overall Officials: Haiyan Si, M.D., Principal Investigator — Chinese PLA General Hospital (301 Military Hospital)
Locations (1):
- Chinese PLA General Hospital (301 Military Hospital), Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No